CLINICAL TRIAL: NCT03497091
Title: Retrospective Review of Amino Acid Formula Use at a Children's Center
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 17.10.US.HCN
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Children Requiring Amino Acid-based Formula Tube Feeding; Enteral Feeding Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enteral Tube fed children: Enteral Formula
  Interventions: Other: Enteral Formula

INTERVENTIONS:
Other: Enteral Formula — Enteral Feeding with an amino acid-based formula

SUMMARY:
This is a retrospective review of data documented in medical records.

DETAILED DESCRIPTION:
This is a retrospective review of data documented in medical records of patients consuming an amino-acid based enteral formula at a pediatric care facility in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Consuming or with a history of consuming an amino acid-based formula

Exclusion Criteria:

* Medical records lacking information on consumption of an amino acid-based formula

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population studied retrospectively will be children in a pediatric feeding center consuming an amino acid-based enteral fomula and meeting the inclusion/ exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Documented indication for formula use | Up to 12 months before formula switch
  Medical diagnosis

SECONDARY OUTCOMES:
Body weight | 12, 6 months prior to formula switch, at formula switch, and 6, 12 months post switch
  Body weight in kilograms
Length/height | 12, 6 months prior to formula switch, at formula switch, and 6, 12 months post switch
  Length or height (based on age) in centimeters
Formula volume consumption | 12, 6 months prior to formula switch, at formula switch, and 6, 12 months post switch
  Average of 7 days
Stool frequency | 12, 6 months prior to formula switch, at formula switch, and 6, 12 months post switch
  Average of 7 days
Stool consistency | 12, 6 months prior to formula switch, at formula switch, and 6, 12 months post switch
  Average of 7 days
Vomiting | 12, 6 months prior to formula switch, at formula switch, and 6, 12 months post switch
  Average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Krysmaru AraujoTorres, MD, Study Director — Société des Produits Nestlé (SPN)
Locations (1):
- Children's Center for Rehabilitation Hospital, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No